CLINICAL TRIAL: NCT04730258
Title: Phase 1b/2 Clinical Study of the Safety, Tolerability, and Pharmacokinetic and Pharmacodynamic Profiles of CFI-400945 as a Single Agent or in Combination With Azacitidine in Patients With AML, MDS or CMML
Brief Title: A Study of CFI-400945 With or Without Azacitidine in Patients With AML, MDS or CMML
Acronym: TWT-202
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Treadwell Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TWT-202
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; AML; MDS; CMML
Keywords: Polo-like kinase 4; PLK4; serine/threonine kinase Polo-like kinase 4; CFI-400945; 945; Polo-Like Kinase 4 inhibitors/antagonists; hematologic malignancies; PLK-4; UHN; University Health Network; Treadwell; Treadwell Therapeutics; Treadwell Tx
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Hematologic Neoplasms | interventions — 2-(3-(4-((2,6-dimethylmorpholino)methyl)styryl)-1H-indazol-6-yl)-5'-methoxyspiro(cyclopropane-1,3'-indolin)-2'-one; Azacitidine

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion for monotherapy and combination arms with azacitidine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1A: Monotherapy escalation and expansion (Experimental): Dose escalation and expansion arm with CFI-400945
  Interventions: Drug: CFI-400945
- 2A: Combination escalation and expansion (Experimental): Dose escalation and expansion arm with CFI-400945 and azacitidine
  Interventions: Drug: CFI-400945; Drug: Azacitidine

INTERVENTIONS:
Drug: CFI-400945 — The starting dose is 32 mg/day for escalation arms and the recommended starting dose for the expansion arms.
  Other Names: CFI-400945 fumarate; 945; 400945
Drug: Azacitidine — Azacitidine will be given at its labeled dose and schedule
  Arms: 2A: Combination escalation and expansion

SUMMARY:
The purpose of this study is to test the safety of an investigational drug called CFI-400945 alone and in combination with azacitidine.

DETAILED DESCRIPTION:
This study will be evaluating the safety and tolerability of CFI-400945 in subjects with Acute Myeloid Leukemia, Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia. The study is designed to build on encouraging data from another study and to obtain further safety, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) data of CFI-400945.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be >18 years of age
2. For Parts 1A and 1B, the following malignancy types will be included:

   1. Relapsed or refractory AML.
   2. MDS, after prior hypomethylating agents.
   3. CMML, with progressive disease/lack of response after hypomethylating agents

   For Parts 1A and 1B, Patients may have relapsed or refractory disease.
3. For Parts 2A and 2B, the following malignancy types will be included:

   1. Relapsed or Refractory AML.
   2. MDS patients should be limited to high risk disease
   3. MDS or CMML should be previously untreated and patients with AML may have relapsed or refractory disease;
4. Have clinically acceptable laboratory screening results (i.e., clinical chemistry, hematology, and urinalysis) within certain limits per protocol.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

1. Patients who have received investigational therapy, radiotherapy, immunotherapy, monoclonal antibodies, or chemotherapy within 14 days or 5 half-lives (whichever is shorter)
2. Allogeneic or autologous transplant for AML with infusion of stem cells within 90 days before Cycle 1 Day 1, or on active immunosuppressive therapy for graft-versus-host disease (GVHD) or GVHD prophylaxis within 2 weeks of Cycle 1 Day 1.
3. Any Grade ≥ 2 persistent non-hematological toxicity related to allogeneic transplant, such as those requiring systemic immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent AEs | 36 months
  The number of subjects who experience an adverse event that was possibly related to study drug
Treatment emergent changes in vital signs | 36 months
  The number of subjects who experience changes in blood pressure, heart rate, respiratory rate, body temperature that was possibly related to study drug.
Treatment emergent changes in clinical laboratory tests | 36 months
  The number of subjects who experience a change in laboratory parameters that was possibly related to study drug.
Treatment emergent changes in physical examinations, ECOG performance status, electrocardiograms (ECGs), echocardiograms and cardiac troponins | 36 months
  The number of subjects who experience changes in physical examinations, performance status, ECG, troponins that were possibly related to study drug.

SECONDARY OUTCOMES:
Composite Complete Remission Rate, CRc (complete remission + complete remission with incomplete blood count recovery + complete remission with incomplete platelet count recovery [CR + CRi + CRp]) | 36 months
  Response rate will be summarized by dose cohort and overall using the percent of patients in patient with AML
Overall response rate (ORR, defined as Complete remission + Marrow CR + Partial remission + Hematologic Improvement (CR + mCR+ PR + HI) | 36 months
  Response rate will be summarized by dose cohort and overall using the percent of patients in patients with MDS, CMML
The pharmacokinetics of CFI-400945 will be assessed through AUC. | 36 months
  Area under the plasma concentration (AUC) versus time curve from time 0 to time of least measurable concentration tabulated by dose group.
To assess the pharmacokinetic profile of CFI-400945 through Cmax. | 36 months
  Cmax will be assessed through the maximum measured plasma concentration occurring at Tmax tabulated by dose group.
To assess the pharmacokinetic profile of CFI-400945 through T1/2. | 36 months
  Elimination half life will be calculated and tabulated by dose group.

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MD, Principal Investigator — The University of Texas MD Anderson Cancer Centre
Locations (9):
- United States (6):
  - City of Hope, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Norton Cancer Institute - Saint Matthews, Louisville, Kentucky
  - New York Presbyterian Weill Cornell Medical Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Centre, Houston, Texas
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Princess Margaret Cancer Center, Toronto, Ontario
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
It is too early to determine whether we will make IPD available - we do not yet have a process written on this. Field will be updated once our policy / process is written.

REFERENCES:
- [Derived] Murphy T, Mason JM, Leber B, Bray MR, Chan SM, Gupta V, Khalaf D, Maze D, McNamara CJ, Schimmer AD, Schuh AC, Sibai H, Trus M, Valiquette D, Martin K, Nguyen L, Li X, Mak TW, Minden MD, Yee KWL. Preclinical characterization and clinical trial of CFI-400945, a polo-like kinase 4 inhibitor, in patients with relapsed/refractory acute myeloid leukemia and higher-risk myelodysplastic neoplasms. Leukemia. 2024 Mar;38(3):502-512. doi: 10.1038/s41375-023-02110-9. Epub 2023 Dec 19. PMID 38114624